CLINICAL TRIAL: NCT04147208
Title: Evaluate the Safety, Tolerability, and Antiviral Activity of GLS4 With Ritonavir in Combination With Entecavir in Comparison With Entecavir Alone in Patients With Chronic HBV Who Are HBeAg Positive
Brief Title: Evaluate the Safety, Tolerability, and Antiviral Activity of GLS4 With Ritonavir in Patients With Chronic HBV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DGLS4-18-002
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Chronic HBV Infection
Keywords: Chronic HBeAg positive HBV Infection
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination group (Experimental): Subjects will receive 96 weeks of GLS4+RTV+ETV.
  Interventions: Drug: GLS4; Drug: RTV; Drug: ETV
- Entecavir monotherapy (Active Comparator): Subjects received 96 weeks of entecavir treatment
  Interventions: Drug: ETV

INTERVENTIONS:
Drug: GLS4 — Administered GLS4 120 mg orally three times daily in fed state
  Other Names: Morphothiadine Mesilate Capsules
  Arms: Combination group
Drug: RTV — Administered RTV 100 mg orally three times daily in fed state
  Other Names: Ritonavir tablet
  Arms: Combination group
Drug: ETV — Administered orally ETV 0.5 mg once daily in fasted state
  Other Names: Entecavir table

SUMMARY:
The experiment is divided into two parts: Part 1 and Part 2.Part 1 was the initial treatment patient and Part 2 was the treated patient.

DETAILED DESCRIPTION:
About 125 subjects were planned to be included and assigned to the experimental group and the control group according to 4:1.At the same time, a liver biopsy group was set up in each part of the population to receive liver biopsy during the screening period and 48 weeks after completion of drug administration, which was used to detect HBV DNA, cccDNA, HBsAg, and evaluate the degree of liver inflammation and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection population
* HBeAg positive
* HBsAg≥250 IU/mL
* No cirrhosis

Exclusion Criteria:

* AST>5×ULN
* Platelet count less than 90E+09/L
* TBil>1.5×ULN
* albumin<35 g/L
* INR>1.5
* AFP>50 ng/mL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
The value of serum HBsAg decreased from baseline | 48 weeks after dosing
  The value of serum HBsAg at 48 weeks of treatment was lowered compared with baseline.

SECONDARY OUTCOMES:
The value of serum HBeAg decreased from baseline | 48 weeks after dosing
  The value of serum HBeAg at 48 weeks of treatment was lowered compared with baseline.
The value of HBV DNA decreased from baseline | 48 weeks after dosing
  The value of HBV DNA at 48 weeks of treatment was lowered compared with baseline.
The value of serum HBsAg decreased from baseline | 24 weeks after dosing
  The value of serum HBsAg at 24 weeks of treatment was lowered compared with baseline.
The value of serum HBeAg decreased from baseline | 24 weeks after dosing
  The value of serum HBeAg at 24 weeks of treatment was lowered compared with baseline.
The value of HBV DNA decreased from baseline | 24 weeks after dosing
  The value of HBV DNA at 24 weeks of treatment was lowered compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: junqi Niu, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (37):
- China (37):
  - Beijing Ditan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The second affiliated hospital of ChongQing medical university, Chongqing, Chongqing Municipality
  - The first affiliated hospital of ChongQing medical university, Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The third affiliated hospital of sun yat-sen university, Guangzhou, Guangdong
  - The first affiliated hospital of Guangxi medical university, Nanning, Guangxi
  - Affiliated hospital of Guizhou medical university, Guiyang, Guizhou
  - Affiliated hospital of ZunYi medical college, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The fourth affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University Science & Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The People's Liberation Army No.81 Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - The Third People's Hospital of Zhenjiang, Zhenjiang, Jiangsu
  - The first hospital of jilin university, Changchun, Jilin
  - The second hospital of jilin university, Changchun, Jilin
  - Qingdao municipal hospital, Qingdao, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Sub-Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai putuo district central hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The second affiliated hospital of air force medical university, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin third central hospital, Tianjing, Tianjing
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Gao Y, Kong F, Gao H, Yi Y, Wu C, Xin Y, Zheng S, Lu J, Han T, Zhao Y, Hu P, Mao X, Xie Q, Zhang J, Hou J, Gao Z, Lian J, Chen L, Shang J, Xie W, Mu M, Jin Z, Wang M, Lin S, Rao H, Yang D, Gong H, Luo L, Chen Y, Zhuang Y, Zhang Y, Gish RG, Tan Y, Zhang J, Niu J. Efficacy and safety of GLS4 with entecavir vs entecavir alone in chronic hepatitis B patients: A multicenter clinical trial. J Infect. 2025 Mar;90(3):106446. doi: 10.1016/j.jinf.2025.106446. Epub 2025 Feb 21. PMID 39988055